CLINICAL TRIAL: NCT00994188
Title: A Clinical Study of the Living-related Renal Transplantation With Restored Kidneys (Interventional Trial)
Brief Title: A Clinical Study of the Living Renal Transplantation With Restored Kidneys Between Family Members
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tokushukai Medical Group (Other)
Responsible Party: Yoshihide Ogawa, Tokyo-West Tokushukai Hospital Transplant Office
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TW062090617KT
Record Dates: First submitted 2009-10-09; First posted 2009-10-14 (Estimated); Last update posted 2009-10-14 (Estimated); Status verified 2009-10

CONDITIONS: Kidney Neoplasm; Kidney Stone; Ureteral Tumor; Ureteral Stricture; Renal Insufficiency
Keywords: Renal tumor; Ureteral tumor; Ureteral stricture; Restored kidney; Renal transplantation; Family members
MeSH Terms: conditions — Kidney Neoplasms; Kidney Calculi; Ureteral Neoplasms; Renal Insufficiency; Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Restored Kidney Transplant Between Family Members — Tumor part of the kidney or ureter and ureteral stricture is surgically removed or repaired and the kidney is restored and transplanted to a family member recipient

SUMMARY:
Approximately 30,000 new patients are introduced into dialysis and about 20,000 of them die every year in Japan. At present, about 300,000 patients are on dialysis and more than 10,000 patients are registered with the Japan Organ Transplant Network (JOTN) with the hope for a renal transplantation. If the renal function is restored by transplantation, the quality of life (QOL) improves and more than 90% are reportedly comeback to their normal life activities and get relieved from the burden of dialysis. Furthermore, it can reduce the dialysis related medical cost by as much as 50%. However, only about 1,000 renal transplantation cases are annually carried out in Japan. Among them, 80-85% are living renal transplantations offered by family members or relatives, and the rest are from deceased donors.

Due to the fact that the number of deceased donors are scarce and only living renal transplantations between the family members or relatives are currently allowed in Japan, the approximate waiting time to receive a renal transplantation is 16 years. For that reason, many patients travel abroad to receive a renal transplantation.

There are reports that total nephrectomies are performed as a treatment for small size (4 cm or less) renal tumors, renal stones, ureteral tumors and ureteral strictures in many cases and that many of these nephrectomized kidneys can be successfully transplanted after surgical restoration with satisfactory results. However, due to the lack of necessary evidence it is currently not allowed in Japan.

Therefore, the investigators planned the present clinical study to evaluate the curative efficacy (renal function, QOL) and safety (side effects, complications or occurrence of renal cancer) of living renal transplantations between family members and relatives with restored donor kidneys after the surgical removal or repairment of a small size (4 cm or less) renal tumor or renal stone, ureteral tumor or ureteral stricture, in order to acquire necessary clinical data for potential enrichment of the renal donor pool in Japan as well as to develop useful medical care for our patients who are on dialysis for many years due to the renal failure.

ELIGIBILITY:
Inclusion Criteria:

A) Recipient:

* Patients who are suffering from renal failure and are willing to receive a restored kidney from a family member
* Patients who are eligible for general anesthesia
* Patients who have given written informed consent to participate in the study

B) Donor:

* Potential donors who are incidentally diagnosed with small renal tumor (size: <4 cm) or renal stone, ureteral tumor or ureteral stricture and have permitted to transplant the kidney to a family member upon its surgical restoration
* Patients who are eligible for general anesthesia
* Patients who have given written informed consent to participate in the study

Exclusion Criteria:

A) Recipient:

* Patients who have infectious disease, hemorrhagic ulcer, or malignant cancer
* Patients who have serious vascular lesions (eg. arteriosclerosis, thromboembolic disease) and are currently on treatment
* Patients who were disapproved by the Institutional Ethics Committee

B) Donor:

* Patients who have tested positive for serious infectious disease (eg. HIV, HBV, or HCV)
* Patients who were diagnosed with malignant lymphoma or sarcoma
* Patients who were on chemotherapy or radiation therapy for renal cancer prior to the nephrectomy
* Patients who were disapproved by the Institutional Ethics Committee

(*) Other inclusion/exclusion criteria defined in the protocol for both recipient and donor may apply.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2009-07; Primary Completion 2014-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Evaluation of curative efficacy (renal function and QOL) and safety (side effects, complications) after renal transplantation with restored kidneys between family members | 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Yoshihide Ogawa, MD, PhD, Principal Investigator — Tokyo-West Tokushukai Hospital
Locations (2):
- Japan (2):
  - Uwajima Tokushukai Hospital, Uwajima, Ehime
  - Tokyo-West Tokushukai Hospital Transplant Office, Akishima, Tokyo